CLINICAL TRIAL: NCT06223828
Title: Azithromycin as Immunomodulation Among Children Hospitalized for Critical Asthma: A Prospective, Open-Label, Non-Randomized, Interventional Study With Parallel Biospecimen Banking
Brief Title: Azithromycin for Critical Asthma - Pediatrics
Acronym: CR-AZI Kids
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-AZI; IRB00410054 (Other: Johns Hopkins University)
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Asthma; Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Children will be enrolled into either a single interventional arm or a parallel standard care arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin Intervention (Experimental): Participants in this arm will receive Azithromycin 10mg/kg/dose (max dose 500mg) once daily for 3 days.
  Interventions: Drug: Azithromycin
- Standard Care (No Intervention): Participants will receive standard care without Azithromycin.

INTERVENTIONS:
Drug: Azithromycin — 10mg/kg/dose (max dose 500mg) once daily for 3 days
  Other Names: Zithromax
  Arms: Azithromycin Intervention

SUMMARY:
The CR-AZI Study will assess the immunomodulatory effects of Azithromycin for pediatric Critical Asthma.

DETAILED DESCRIPTION:
Azithromycin (AZI), a macrolide antibiotic, has been applied for adult and pediatric respiratory pathology to alter immune system response.1 For pediatric critical asthma (CA), a term used to describe a critically ill child hospitalized with an asthma exacerbation requiring an intensive care unit (PICU) hospitalization, the investigator's prior research has revealed 1 in 10 will receive AZI.2 Yet, the application of AZI in this setting is poorly studied nor is clear if, and to what degree AZI alters the immune response in conjunction with systemic corticosteroids traditionally applied in CA.

In this proposal, the investigators aim to characterize a respiratory epithelial inflammatory biomarker, periostin, among children with CA with and without exposure to AZI. The investigators hypothesize children receiving AZI will have lower periostin levels. As a secondary analysis, the investigators will describe the rates of adverse events related to AZI (previously not done) and explore differences in clinical and physiologic CA efficacy markers.

ELIGIBILITY:
Inclusion criteria

* Age 3-17 years
* Admission to the PICU
* Primary diagnosis of critical asthma
* Prescription for continuous inhaled beta-agonist therapy and/or intravenous (IV) beta-agonist therapy
* Prescription for intravenous systemic corticosteroids

Exclusion criteria

* Critical Congenital Heart Disease Unrepaired
* Tracheostomy Dependence at Admission
* Ongoing Exposure to Azithromycin or Macrolide Antibiotics for any indication
* Past Medical History of Prolonged QT Syndrome or Arrhythmias
* Concomitant respiratory pathology including Acute Chest Syndrome, Interstitial Lung Disease, Cystic Fibrosis, and pulmonary hypertension

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma Periostin Levels and Degree of Change (e.g., Slope) - Primary Physiologic Efficacy Endpoint | 24 hours, 48 hours, and 72-hours following enrollment
  ng/dL
Drug-related adverse event rate (Primary Safety Endpoint) | During hospitalization, approximately 3 days
  cumulative incidence rate

SECONDARY OUTCOMES:
Length of Stay (Secondary Clinical Efficacy Endpoint) | During hospitalization, approximately 3 days
  Measured in Days, from Hospitalization in ICU through Discharge from ICU
Duration of continuous albuterol (Secondary Clinical Efficacy Endpoint) | During hospitalization, approximately 3 days
  Measured in Hours from ICU hospitalization through discharge
Composite use of adjunct asthma treatments (Secondary Clinical Efficacy Endpoint) | During hospitalization, approximately 3 days
  Cumulative Frequency of Exposure, from ICU Hospitalization through ICU discharge
Transcutaneous carbon dioxide levels (Secondary physiologic efficacy Endpoint) | Enrollment, Day 1, Day 2, Day 3, at ICU Discharge
  Measured in mmHg of Carbon Dioxide, peak values measured daily at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A Sochet, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share with other researchers.